CLINICAL TRIAL: NCT00304590
Title: A Phase 2 Study of XL999 in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: Study of XL999 in Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to cardiac toxicities in the subjects
Sponsor: Symphony Evolution, Inc. (Industry)
Responsible Party: Charles W. Finn, PhD, President and CEO, Symphony Evolution, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL999-203
Record Dates: First submitted 2006-03-16; First posted 2006-03-20 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: XL999 — Treatment consisted of 8 weekly infusions of 2.4 mg/kg of XL999 with each infusion given over 4 hours, unless drug-related toxicity required a dosing delay or adjustment. In the absence of progressive disease and unacceptable toxicity, subjects may have received XL999 treatment weekly for up to 1 year on this study.

SUMMARY:
This clinical study is being conducted at multiple sites to determine the activity, safety, and tolerability of XL999 when given weekly to patients with relapsed or refractory multiple myeloma. XL999 is a small molecule inhibitor of cellular factors including VEGFR, PDGFR, and FGFR that may be involved in multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with a diagnosis of MM based on bone marrow aspirate and biopsy with ≥10% plasma cells (or biopsy of a tissue with monoclonal plasma cells), M protein level in the serum or urine, and evidence of end organ or tissue impairment (hypercalcemia, renal insufficiency, anemia, or lytic bone lesions), as defined by The International Myeloma Working Group Criteria (2003), at initial diagnosis (before initiation of chemotherapy)
* Measurable disease defined as serum and/or urine M component by electrophoresis
* Refractory to or relapsed after 2 prior treatment regimens (chemotherapy, biologic or hematopoietic stem cell transplantation)
* Concurrent therapy with a bisphosphonate is acceptable
* ECOG performance status of 0 or 1
* Life expectancy ≥3 months
* Adequate liver function
* No other malignancies within 5 years
* Signed informed consent

Exclusion Criteria:

* Nonsecretory myeloma, monoclonal gammopathy of uncertain significance (MGUS), or smoldering myeloma
* Anticancer therapy including chemotherapeutic, biologic, or investigational agents, including dexamethasone, within 30 days of XL999 treatment
* Hematopoietic stem cell transplantation within the previous 6 weeks
* Radiation to ≥33% of bone marrow within 30 days of XL999 treatment
* Subject has not recovered to grade ≤1 or to within 10% of baseline from adverse events due to investigational or chemotherapeutic drugs that were administered >30 prior to study enrollment
* Uncontrolled and/or intercurrent illness
* Pregnant or breastfeeding females
* Known HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-02; Primary Completion 2006-12 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Response rate | Inclusion of subject until disease progression
Safety and tolerability | Inclusion until 30 days post last treatment

SECONDARY OUTCOMES:
Duration of response | Inclusion until disease progression
Progression-free survival | Inclusion until disease progression
Overall survival | Inclusion until 180-day Follow-up or death

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Bui, MD, Study Director — Exelixis
Locations (3):
- United States (3):
  - UCLA Oncology-Hematology Associates, Ltd., Los Angeles, California
  - University of Chicago, Chicago, Illinois
  - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois